CLINICAL TRIAL: NCT00323570
Title: A Multi-center, Randomized, Double-blind, Parallel Group, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Activated Recombinant Factor VII (rFVIIa/NovoSeven®/ NiaStase®) in the Treatment of Refractory Bleeding in Severely Injured Trauma Patients
Brief Title: Evaluation of Recombinant Factor VIIa in Patients With Severe Bleeding Due to Trauma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Public Access to Clinical Trials, Novo Nordisk A/S
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7TRAUMA-1648
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-03

CONDITIONS: Acquired Bleeding Disorder; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: activated recombinant human factor VII

SUMMARY:
This trial is conducted in the United States of America (USA). The purpose of this study is to evaluate the treatment of Recombinant Faction VIIa in Patients with Severe Bleeding Due to Trauma

Please note that this trial and trial F7TRAUMA-1711 (NCT00184548) have been merged.

ELIGIBILITY:
Inclusion Criteria:

* Trauma injury (blunt and/or penetrating) with evidence of active torso hemorrhage refectory to standard treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Mortality and Morbidity | through day 30

SECONDARY OUTCOMES:
All cause mortality
Hospital-free days
Number of transfusion units
Days free of renal replacement therapy
ICU-free days
Days free of ventilator support

CONTACTS AND LOCATIONS:
Overall Officials: Bartholomew Tortella, MD, Study Director — Novo Nordisk A/S
Locations (40):
- United States (40):
  - Novo Nordisk Clinical Trial Call Center, Phoenix, Arizona
  - Novo Nordisk Clinical Trial Call Center, Los Angeles, California
  - Novo Nordisk Clinical Trial Call Center, Sacramento, California
  - Novo Nordisk Clinical Trial Call Center, Colorado Springs, Colorado
  - Novo Nordisk Clinical Trial Call Center, Washington D.C., District of Columbia
  - Novo Nordisk Clinical Trial Call Center, Gainesville, Florida
  - Novo Nordisk Clinical Trial Call Center, Jacksonville, Florida
  - Novo Nordisk Clinical Trial Call Center, Miami, Florida
  - Novo Nordisk Clinical Trial Call Center, Chicago, Illinois
  - Novo Nordisk Clinical Trial Call Center, Maywood, Illinois
  - Novo Nordisk Clinical Trial Call Center, Indianapolis, Indiana
  - Novo Nordisk Clinical Trial Call Center, Louisville, Kentucky
  - Novo Nordisk Clinical Trial Call Center, Portland, Maine
  - Novo Nordisk Clinical Trial Call Center, Baltimore, Maryland
  - Novo Nordisk Clinical Trial Call Center, Boston, Massachusetts
  - Novo Nordisk Clinical Trial Call Center, Detroit, Michigan
  - Novo Nordisk Clinical Trial Call Center, Springfield, Missouri
  - Novo Nordisk Clinical Trial Call Center, St Louis, Missouri
  - Novo Nordisk Clinical Trial Call Center, Las Vegas, Nevada
  - Novo Nordisk Clinical Trial Call Center, Camden, New Jersey
  - Novo Nordisk Clinical Trial Call Center, Brooklyn, New York
  - Novo Nordisk Clinical Trial Call Center, The Bronx, New York
  - Novo Nordisk Clinical Trial Call Center, Greenville, North Carolina
  - Novo Nordisk Clinical Trial Call Center, Winston-Salem, North Carolina
  - Novo Nordisk Clinical Trial Call Center, Akron, Ohio
  - Novo Nordisk Clinical Trial Call Center, Cleveland, Ohio
  - Novo Nordisk Clinical Trial Call Center, Columbus, Ohio
  - Novo Nordisk Clinical Trial Call Center, Oklahoma City, Oklahoma
  - Novo Nordisk Clinical Trial Call Center, Portland, Oregon
  - Novo Nordisk Clinical Trial Call Center, Allentown, Pennsylvania
  - Novo Nordisk Clinical Trial Call Center, Philadelphia, Pennsylvania
  - Novo Nordisk Clinical Trial Call Center, Pittsburgh, Pennsylvania
  - Novo Nordisk Clinical Trial Call Center, Providence, Rhode Island
  - Novo Nordisk Clinical Trial Call Center, Memphis, Tennessee
  - Novo Nordisk Clinical Trial Call Center, Nashville, Tennessee
  - Novo Nordisk Clinical Trial Call Center, Fort Sam Houston, Texas
  - Novo Nordisk Clinical Trial Call Center, Lackland Air Force Base, Texas
  - Novo Nordisk Clinical Trial Call Center, San Antonio, Texas
  - Novo Nordisk Clinical Trial Call Center, Salt Lake City, Utah
  - Novo Nordisk Clinical Trial Call Center, Madison, Wisconsin

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com